CLINICAL TRIAL: NCT04754997
Title: The Effect of Exercise Training on Pain, Physical Activity and Quality of Life in Pediatric Hemophilia Patients
Brief Title: Effect of Exercise in Pediatric Hemophilia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/116
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Hemophilia A, Severe; Hemophilia Arthropathy
Keywords: Hemophilia; Factor VIII; Closed chain exercise; Knee
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Participants were divided in three groups. Two groups will get two different intervention. One group will be the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): This group will not take any exercise intervention.
- Traditional exercise training group (Active Comparator): This group will get traditional therapy that is include range of motion exercises and resistance exercise training.
  Interventions: Other: Traditional exercise training
- Specific exercise training group (Experimental): This group will get a specific programme that combinated with closed kinetic chain exercises and core exercises training
  Interventions: Other: Specific exercise training

INTERVENTIONS:
Other: Traditional exercise training — The therapy program will planned for 12 weeks and the sessions will be performed in 45 minutes (min) for 2 days a week. The lower extremity range of motion exercise and strengthening exercises will be applied on the mat 10 repetition. The number of repetitions and type of exercises will be changed every 3 weeks.
  Arms: Traditional exercise training group
Other: Specific exercise training — The therapy program will planned for 12 weeks and the sessions will be performed in 45 minutes (min) for 2 days a week. Exercise training consists of lower extremity closed kinetic chain exercises and core exercises. The type of exercise changes every 3 weeks.
  Arms: Specific exercise training group

SUMMARY:
This study investigates the effect of exercise training on pain, physical activity and quality of life in pediatric hemophilia patients.

DETAILED DESCRIPTION:
Hemophilia is a congenital X-linked recessive disease characterized by the lack or absence of clotting factors in the blood. Male individuals with problems in the X chromosome are affected, females are carriers. There are two common types, factor VIII (Hemophilia A) and factor IX (Hemophilia B), and the percentage of the exposed factor in circulation determines the degree of hemophilia disease (<1% severe, 1-5% moderate,> 20% mild). The most common clinical symptoms in hemophilia are intra-articular and intramuscular spontaneous bleeding, a history of bleeding that lasts longer than expected after trauma, hemarthrosis and hematomas after crawling or walking in children with moderate or severe hemophilia. Pain, swelling, redness, temperature increase and limitation of movement occur in the bleeding joint. Bleeding into the joint space causes inflammation in the synovial membrane and synovitis occurs. With chronic synovitis, the synovial membrane thickens. Degeneration of the joint cartilage and narrowing of the joint space occurs. Hemarthroses constitute 70-80% of bleeding findings. The most common bleeding joints are knee joints with a rate of 45%. Besides pharmacological treatment for joint and muscle bleeding, the most suitable option is exercise therapy.

The aim of our study is to examine the effect of exercise agitation on pain, physical activity and quality of life in pediatric hemophilia patients. The results of the study indicate that the exercise protocol developed for the lower extremity in pediatric hemophilia patients will have a positive effect on pain, physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hemophilia (Hemophilia A) by a hematologist
* Hemophilia is moderate or severe, without spontaneous bleeding complaints
* Having a history of bleeding in the knee joint
* Not doing any regular exercise
* Willing to continue working and will not start other treatment during the study
* Patients whose parents were informed about the study and whose consent form was obtained

Exclusion Criteria:

* Those who have undergone another surgery (joint debridement, fracture, knee replacement) that will affect lower extremity function
* Those with neurological disease or any sensory loss or peripheral nerve injury that may affect functional performance and balance

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Hemophilia a disease is an X-linked recessive disease. Therefore, girls become carriers and do not show muscle joint problems.
Enrollment: 30 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
The Pain | through of the study, average 12 weeks
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Functional ambulatory mobility | through of the study, average 12 weeks
  Time Up and Go test will used to determine ambulatory mobility. Time up and go test required documenting the time in seconds that subjects required to: "rise from a standard arm chair, walk to a line on the floor 3 meters away, turn, return, and sit down again." If relapsed time score is increased, that is mean mobility function will worse.
Functional exercise capacity | through of the study, average 12 weeks
  Two minutes walk test will used to determine physical activity. 2-minute walk test (2MWT) is classified to represent the most suitable method to assess the submaximal level of functional exercise capacity in children. This test measures the distance that a patient or participant quickly walk on a flat, hard surface in a period of 2 minutes.If the covered distance is increased, that is mean functional capacity will worse.
Lower extremity functional strength test | through of the study, average 12 weeks
  Sit to stand test will used to determine physical activity. The sit-to-stand test measures time needed to complete three consecutive sit-to-stand cycles as quickly as possible. The higher the rate of three-repetition sit-to-stand (repetitions per second), the more strength a children has.
The quality of Life | through of the study, average 12 weeks
  The Children's Quality of Life Scale ( PedsQL) will used to determine to quality of life level. The quality of life scale for children questions the last month of children and adolescents. It is a 5-point Likert-type scale with never 100 points, rarely 75 points, sometimes 50 points, often 25 points and always 0 points. The total score is obtained by dividing the scores obtained from the scale by the number of filled items. The higher the total score, the better the quality of life.

SECONDARY OUTCOMES:
Knee Proprioception | through of the study, average 12 weeks
  Electro goniometer measurement will used to determine knee proprioception
Joint Health | through of the study, average 12 weeks
  Hemophilia Joint Health Scale will used to determine bilaterally knee, elbow and ankle joint health. Total score of the scale is 124 point. The higher score of the scale, the more deficit joints have.
Functional Independence | through of the study, average 12 weeks
  Functional Independence Score in Hemophilia (FISH) will used to functional independence. FISH is based on observing the performance of daily life activities. Patients are assessed for their ability to perform eight tasks, divided into three categories: self-care (eating, grooming, bathing and dressing), transfers (chair and squatting) and mobility (walking, going up stairs and running).The scores achieved in each task are summed giving a total from 8 to 32 points with 32 indicating the highest level of functional independence
Static Balance | through of the study, average 12 weeks
  Stand on one leg test was used assess static balance

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Vulpen LFD, Holstein K, Martinoli C. Joint disease in haemophilia: Pathophysiology, pain and imaging. Haemophilia. 2018 May;24 Suppl 6:44-49. doi: 10.1111/hae.13449. PMID 29878659
- [Background] Wagner B, Kruger S, Hilberg T, Ay C, Hasenoehrl T, Huber DF, Crevenna R. The effect of resistance exercise on strength and safety outcome for people with haemophilia: A systematic review. Haemophilia. 2020 Mar;26(2):200-215. doi: 10.1111/hae.13938. Epub 2020 Feb 24. PMID 32091659
- [Background] Siqueira TC, Dominski FH, Andrade A. Effects of exercise in people with haemophilia: An umbrella review of systematic reviews and meta-analyses. Haemophilia. 2019 Nov;25(6):928-937. doi: 10.1111/hae.13868. Epub 2019 Oct 30. PMID 31667968
- [Background] Souza JC, Simoes HG, Campbell CS, Pontes FL, Boullosa DA, Prestes J. Haemophilia and exercise. Int J Sports Med. 2012 Feb;33(2):83-8. doi: 10.1055/s-0031-1286292. Epub 2011 Nov 17. PMID 22095329